CLINICAL TRIAL: NCT06301490
Title: The Effect of Myofascial Release in Patients With Subacromial Impingement Syndrome Randomized Controlled Trial
Brief Title: The Effect of Myofascial Release in Patients With Subacromial Impingement Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taif University (Other)
Responsible Party: Principal Investigator, Adel Muawidh Alqarafi, Principal Investigator, Taif University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Taif university
Record Dates: First submitted 2024-03-02; First posted 2024-03-08 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Subacromial Impingement Syndrome
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): 18 participants will have strengthening exercises, rang of motion exercises and ice application for 10 mins
- experimental group (Experimental): 18 participants will have strengthening exercises, rang of motion exercises and ice application for 10 mins, with adding Myofascial Release
  Interventions: Other: Myofascial Release

INTERVENTIONS:
Other: Myofascial Release — Myofascial release is a popular hands-on method manual therapy technique that uses carefully guided low load, long duration mechanical pressures to modify the myofascial complex (directly or indirectly), with the goal of restoring appropriate length, decreasing discomfort, and improving range of motion, muscle recovery, and physical performance in healthy persons.
  Arms: experimental group

SUMMARY:
BACKGROUND: Shoulder pain has been reported to be the third most common musculoskeletal presentation in primary care, after low back pain and knee pain. The prognosis for those presenting with musculoskeletal shoulder pain varies greatly amongst individuals, with 50% of people reporting symptoms 6 months after presenting in primary healthcare. Functional limitations, in addition to pain, are widespread and can interfere with job, hobbies, social, and sporting activities. They may also relate to psychological discomfort and a lower quality of life. Continuous computer uses without a break, awkward postures, and the duration and frequency of laptop use have all been identified as risk factors for musculoskeletal diseases. The most prevalent cause, accounting for 70% of cases, is rotator cuff dysfunction. Rotator cuff disorders are frequently associated with short and long-term impairment and discomfort, with approximately fifty percent of patients experiencing pain or functional restrictions for up to two years. The majority of shoulder pain concerns are treated in primary care by physiotherapists and general practitioners. Myofascial release is a common hands-on method manual therapy technique that uses carefully guided low load, long duration mechanical pressures to modify the myofascial complex with promising results in improving functional level.

OBJECTIVE: The purpose of this study is to investigate the effect of myofascial release in patient with rotator cuff tendinopathy.

METHOD: The design of this study is a double blinded Randomize control trail. Forty-two participants will be divided into one of two groups, group one will have strengthening exercises, range of motion exercise, and ice application, group two will perform the same exercises with ice application plus myofascial release. Patient will be followed for one month, two session per week and the session duration will be 30-45 mins. Assessment and re-assessment will be done by independent physical therapist. All patients will be assessed by using quick DASH, VAS, ROM, and Kessler psychological distress scale.

ELIGIBILITY:
Inclusion Criteria:

1. are aged between 20-60 years old,
2. have one or more than one positive finding in one of the following categories: (1) painful arc of movement during flexion or abduction; (2) Neer (sensitivity 0.78, specificity 0.58) or Kennedy-Hawkins (sensitivity 0.74, specificity 0.57) impingement signs[28]; and (3) pain during resisted external rotation, abduction or empty can test (sensitivity 0.69, specificity 0.62).[29] A combination of positive results to these clinical tests has values ≥ 0.74 for sensitivity and specificity for SIS.

Exclusion Criteria:

1. have a history of glenohumeral luxation in the last 12 months or any fracture to the shoulder girdle.
2. have a shoulder pain reproduced by cervical movements. had a previous shoulder surgery, adhesive capsulitis, defined as loss of passive shoulder ROM greater than 50%, and
3. have a clinical sign of full-thickness tears of any rotator cuff muscles identified by lag signs [30]: drop sign (sensitivity 0.73, specificity 0.77), external rotation sign (sensitivity 0.46, specificity 0.94) and internal rotation sign (sensitivity 1.00, specificity 0.84).

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2024-01-11 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-03-02 (Actual)

PRIMARY OUTCOMES:
pain intensity | one month
  The pain intensity will be assessed using the visual analogue scale (VAS) which assess pain from 0 (no pain) to 10 (most severe pain) and has good reliability and validity
disability | one month
  The disability will be assessed using Quick DASH. The Arabic Q-DASH questionnaire consist of eleven questions that measures the disability of upper extremity, ranges from 0-100 a higher score indicates a higher disability, and it is a reliable and valid upper extremity outcome measure for assessing patients with various upper extremity disorders

SECONDARY OUTCOMES:
rang of motion | one month
  ROM will be measured in standing position for shoulder flexion, extension, and abduction, supine position for internal rotation, and external rotation with a two-arm standard goniometer with a good reliability
psychological distress, and health-related quality of life (HRQoL) | one month
  HRQoL will be assessed using Kessler psychological distress scale, the questionnaire consists of ten questions, and scoring from 10-50 while 10 means likely will and 50 means likely to have a sever disorder, and it is valid and reliable

CONTACTS AND LOCATIONS:
Locations (1):
- Taif University, Ta'if, Mecca Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided